CLINICAL TRIAL: NCT00005054
Title: Phase II Trial of Temodal 4 Hourly in Progressive Breast Cancer
Brief Title: Temozolomide in Treating Women With Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067649; CHNT-H98-198-50; EU-99047
Record Dates: First submitted 2000-04-06; First posted 2004-06-08 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-01

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating women who have advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the therapeutic activity of temozolomide in terms of tumor response, progression free and overall survival in women with advanced breast cancer. II. Assess the extent of ATase depletion and DNA methylation in the peripheral blood of these patients undergoing this regimen and investigate the relationship between these parameters and tumor response.

OUTLINE: Patients receive oral temozolomide every 4 hours for a total of 5 doses. Treatment continues every 28 days for a minimum of 2 courses and a maximum of 1 year in the absence of unacceptable toxicity or disease progression. Patients are followed at 30 days, and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced carcinoma of the breast with documented progression on first line chemotherapy Measurable disease Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) AST no greater than 3 times ULN Alkaline phosphatase less than 2 times ULN unless arising from bone Renal: Creatinine less than 1.5 times ULN Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other clinically significant disease that would interfere with study evaluations No uncontrolled vomiting that would preclude administration of oral medications HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy and recovered Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: Recovered from prior radiotherapy Surgery: Recovered from prior surgery Other: No other concurrent experimental drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-05

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Howell, MD, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital N.H.S. Trust, Manchester, England, United Kingdom